CLINICAL TRIAL: NCT00332774
Title: A 3-Month Clinical Safety Comparison of Nevanac 0.1% to Acular LS 0.4% and Vehicle Following Cataract Surgery
Brief Title: Nevanac 3-Month Safety Study With QID Dosing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-20
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Postoperative Period

ARMS (3):
- Nevanac (Experimental)
  Interventions: Drug: Nepafenac ophthalmic solution 0.1%
- Acular (Active Comparator)
  Interventions: Drug: Ketorolac Tromethamine ophthalmic solution 0.4%
- Vehicle (Placebo Comparator)
  Interventions: Other: Nepafenac ophthalmic suspension vehicle

INTERVENTIONS:
Drug: Nepafenac ophthalmic solution 0.1% — 1 drop 4 times daily for 90 days
  Arms: Nevanac
Drug: Ketorolac Tromethamine ophthalmic solution 0.4% — 1 drop 4 times daily for 90 days
  Arms: Acular
Other: Nepafenac ophthalmic suspension vehicle
  Other Names: 1 drop 4 times daily for 14 days after surgery
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine the safety of Nevanac 0.1% compared to Acular LS 0.4% and Vehicle in patients treated before cataract surgery and for approximately 90 days following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any race or sex ages 10 years or older undergoing cataract extraction with planned implantation of a posterior chamber intraocular lens.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 10
* Other protocol-defined exclusion criteria may apply

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2006-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Macular thickness

SECONDARY OUTCOMES:
contrast sensitivity, corneal staining, VA, IOP, slit-lamp parameters, fundus parameters

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lane, Study Director — Medical Monitor
Locations (1):
- Contact Alcon for Trial Locations, Fort Worth, Texas, United States